CLINICAL TRIAL: NCT02745444
Title: Prevention of Acute Kidney Injury - Molecular Mechanisms of Dietary Pre-conditioning in Human
Acronym: CR_LSP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Cologne (Other)
Responsible Party: Principal Investigator, Volker Burst, MD, University of Cologne
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: CR_LSP
Record Dates: First submitted 2016-03-29; First posted 2016-04-20 (Estimated); Last update posted 2021-09-29 (Actual); Status verified 2021-09

CONDITIONS: Chronic Kidney Disease
Keywords: Living kidney transplantation; Chronic kidney disease; Acute kidney injury
MeSH Terms: conditions — Renal Insufficiency, Chronic; Acute Kidney Injury | interventions — Diet, Protein-Restricted

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- low-calorie formula diet (Other): Donor taking low-calorie formula diet, 50% of basal energy rate, individually calculated with Mifflin-St. Jeor formula.
  Interventions: Dietary Supplement: low-calorie formula diet
- no diet (No Intervention): Donor ingesting food as usual.
- protein-restricted diet (Other): Donor taking protein-restricted diet according to diet plans of clinical dietetics of University Hospital of Cologne, with unchanged calorie supply, individually calculated with Mifflin-St. Jeor formula.
  Interventions: Dietary Supplement: protein-restricted diet
- Normal protein supply (No Intervention): Donor taking same dishes as protein-restricted diet group but with customary protein levels, with unchanged calorie supply.

INTERVENTIONS:
Dietary Supplement: low-calorie formula diet
  Arms: low-calorie formula diet
Dietary Supplement: protein-restricted diet
  Arms: protein-restricted diet

SUMMARY:
The key objective of this pilot study is to assess the molecular mechanisms of renal pre-conditioning by a one-week low-calorie diet in humans.

The protective effect of the low-calorie diet and also of the protein-restriction in donor on transplant qualities and functions in receptor will also be investigated.

Analysis of transcriptome, lipidome, metabolome, epigenome, proteome und phosphoproteome through tissue samples as well as blood samples for comparison of low-calorie diet, protein-restriction and no-diet groups.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years
* Competent patients
* Planned living kidney transplantation
* Provision of informed consent
* BMI ≥ 18,5 kg/m²

Exclusion Criteria:

* None

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2015-04 (Actual); Primary Completion 2019-05-17 (Actual); Study Completion 2020-05 (Actual)

PRIMARY OUTCOMES:
Number of differentially regulated genes on a transcriptomic level | up to 1 year upon receipt of the last tissue sample
  Identification of relevant difference with regard to transcriptome in kidney tissue between patients with low-calorie diet and and no-diet patients.
Number of differentially regulated genes on a lipidome level | up to 2 years upon receipt of the last tissue sample
  Identification of relevant difference with regard to lipidome in kidney tissue between patients with low-calorie diet and and no-diet patients.
Number of differentially regulated genes on a metabolome level | up to 2 years upon receipt of the last tissue sample
  Identification of relevant difference with regard to metabolome in kidney tissue between patients with low-calorie diet and and no-diet patients.
Number of differentially regulated genes on a epigenome level | up to 2 years upon receipt of the last tissue sample
  Identification of relevant difference with regard to epigenome in kidney tissue between patients with low-calorie diet and and no-diet patients.
Number of differentially regulated genes on a proteome level | up to 1 year upon receipt of the last tissue sample
  Identification of relevant difference with regard to proteome in kidney tissue between patients with low-calorie diet and and no-diet patients.
Number of differentially regulated genes on a phosphoproteome level | up to 2 years upon receipt of the last tissue sample
  Identification of relevant difference with regard to phosphoproteome in kidney tissue between patients with low-calorie diet and and no-diet patients.

SECONDARY OUTCOMES:
Change of NGAL in urine | Preoperative from donor and receptor; 6h, 12h and 24h after renal transplantation from receptor.
  Change of NGAL in urine, marker for kidney damage measured preoperative in donor and receptor.
Cystatin C | Preoperative and up until 7 days after renal transplantation from receptor.
  Marker for kidney damage measured preoperative and daily until Day 7 postoperative in receptor.
Occurrence of acute kidney injury | Assessed up to approx. 30 days from date of renal transplantation until date of discharge, which is the end of observation.
  Occurrence of acute kidney injury according to KDIGO I, II, III in receptor.
Maximum postoperative serum creatinine | Assessed up to approx. 30 days from date of renal transplantation until date of discharge, which is the end of observation.
  Maximum postoperative serum creatinine of receptor during hospital stay.

CONTACTS AND LOCATIONS:
Overall Officials: Volker Burst, MD, Principal Investigator — Principal Investigator
Locations (1):
- University Hospital of Cologne, Cologne, Germany

IPD SHARING:
Plan to Share IPD: Undecided